CLINICAL TRIAL: NCT00685035
Title: Comparison of Sine Waveform High Frequency Chest Wall Oscillation Using Different Settings in Cystic Fibrosis
Brief Title: Comparison of Airway Clearance Therapy in Cystic Fibrosis Using the Same VEST Therapy Device But With Different Settings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0802M26441
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Cystic Fibrosis
Keywords: high frequency chest wall oscillation, cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HFCWC with higher pressure/variable frequency settings (Active Comparator): Half patients randomly assigned to perform HFCWC therapy first with a higher pressure/variable frequency protocol. This entailed performing a 30 minute session with pressure of 10 and 5 minutes each at frequencies of 8,9, and 10 Hz followed by pressure of 6 and 5 minutes each at frequencies of 18, 19, and 20 Hz. This group subsequently crossed-over to the lower-pressure/mid-frequency HFCWC protocol after a washout period of 2 days. This entailed performing a HFCWC session using a pressure of 5 and frequency of 12 Hz for the entire 30 minute session. The other half of subjects were randomly assigned to perform the lower-pressure/mid-frequency protocol first followed by the higher pressure/mixed-frequency after the 2 day washout period
  Interventions: Device: HFCWC with higher pressure/variable-frequency settings; Device: HFCWC with lower pressure/mid-frequency settings
- HFCWC with lower pressure/mid-frequency settings (Active Comparator): lower-pressure/mid-frequency protocol first followed by the higher pressure/mixed-frequency
  Interventions: Device: HFCWC with higher pressure/variable-frequency settings; Device: HFCWC with lower pressure/mid-frequency settings

INTERVENTIONS:
Device: HFCWC with higher pressure/variable-frequency settings — Randomized crossover trial of airway clearance therapy comparing sine wave HFCWO with high pressures and variable frequency (pressure 10, frequencies 8,9,10 and pressure 6, frequencies 18,19,20) to low pressure and mid frequency (pressure 5, frequency 12). Subjects will have 2-day washout between airway clearance sessions. All sputum collected during sessions.
  Other Names: High frequency chest wall oscillation
Device: HFCWC with lower pressure/mid-frequency settings — Subjects will perform pulmonary function tests prior to and following each airway clearance therapy. All sputum produced during, and for 15 minutes following airway clearance therapy will be collected. Subjects will complete a questionnaire addressing the comfort of therapy upon completion of the session.
  Other Names: high frequency chest wall oscillation

SUMMARY:
Our primary hypothesis is that airway clearance therapy with sine waveform HFCWO using higher inflation pressures combined with both low and high oscillator frequencies will result in greater sputum production compared to sine waveform HFCWO with lower inflation pressures and mid-frequency oscillations.

DETAILED DESCRIPTION:
Patients with cystic fibrosis (CF) perform daily airway clearance therapy to facilitate removal of secretions from their airways. Many different techniques are available to achieve this and there is currently no consensus as to which form of therapy is most effective. High frequency chest wall oscillation (HFCWO) is used by CF patients throughout the United States and abroad. To perform this therapy, the patient wears a vest which fits over the entire torso and is connected to an air compressor. The compressor generates oscillating air pulses that are transmitted to the lungs, thereby mobilizing secretions. The most commonly used device is The Vest™ Airway Clearance System, (Hill-Rom Inc, St Paul, MN). Adjustment of the inflation pressure and frequency of oscillations affects the volume of displaced air and flow of air measured at the mouth of the patient. Previous studies indicate this form of therapy is as effective as more traditional and cumbersome forms of therapy. However, it is unclear which inflation pressures and oscillator frequencies provide optimal airway clearance. Some studies of sine waveform HFCWO reported the largest volume of air displacement and highest air flow measured at the mouth when using a combination of high inflation pressures with either low (7 - 10 Hz) or high frequencies (18 - 20 Hz), but most CF centers in the United States use HFCWO with lower pressures combined with mid-range frequencies (10 - 14 Hz). Furthermore, there are no previous studies assessing the affect of sine waveform HFCWO settings on sputum production. As a result, there is no consensus on which pressure and frequency settings are most efficacious for CF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CF established by sweat chloride > 60 mmol/L.
2. Age older than 18 years.
3. History of chronic daily sputum production.
4. Currently on a home therapeutic regimen that includes some form of airway clearance performed with a HFCWO device at least once daily that also includes concomitant use of an inhaled mucolytic and inhaled bronchodilator.
5. FVC and FEV1 > 40%-predicted, and with stable lung function (no greater than a 10% variation in lung function parameters over the preceding 3 months).
6. Evaluated at the University of Minnesota CF Center 3 or more times in the preceding 12 months.

Exclusion criteria:

1. Hospitalization for CF pulmonary complications in the 2 months preceding enrollment.
2. Hemoptysis > 60 cc in a single episode in the 4 weeks preceding enrollment.
3. Chest pain requiring use of narcotic for pain control.
4. Current participation in another clinical trial.
5. Use of intravenous antibiotics for CF respiratory complications in the 2 months preceding enrollment.
6. No prior experience using HFCWO devices for airway clearance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert R Kempainen, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Kempainen RR, Milla C, Dunitz J, Savik K, Hazelwood A, Williams C, Rubin BK, Billings JL. Comparison of settings used for high-frequency chest-wall compression in cystic fibrosis. Respir Care. 2010 Jun;55(6):695-701. PMID 20507651

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potentially eligible patients were identified by query of the Minnesota CF database based on age and FEV1. This list was then reviewed and patients who met additional eligibility requirements were contacted by phone or recruited during a clinic visit by one of the study investigators. Enrollment was completed between 6/1/08 and 10/31/08.
Groups:
- Higher Pressure/Variable-freq, Then Lower Pressure/Mid-freq: HFCWC therapy first with a higher pressure/variable frequency protocol (1st Intervention). After a washout period of 2 days, this group subsequently crossed-over to the lower-pressure/mid-frequency HFCWC protocol (2nd Intervention).
- Lower Pressure/Mid-freq, Then Higher Pressure/Variable-freq: HFCWC therapy first with a lower pressure/mid-frequency protocol (1st Intervention). After a washout period of 2 days, this group subsequently crossed-over to the higher-pressure/variable frequency HFCWC protocol (2nd Intervention).
Period: Period 1: First Intervention: 30 Minutes
Arm/Group | Higher Pressure/Variable-freq, Then Lower Pressure/Mid-freq | Lower Pressure/Mid-freq, Then Higher Pressure/Variable-freq
Started | 9 | 8
Completed | 8 | 8
Not Completed | 1 | 0
Not completed — Pulmonary lab plethysmography malfunctio | 1 | 0
Period: Period 2: 2-day Washout
Arm/Group | Higher Pressure/Variable-freq, Then Lower Pressure/Mid-freq | Lower Pressure/Mid-freq, Then Higher Pressure/Variable-freq
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Period 3: 2nd Intervention
Arm/Group | Higher Pressure/Variable-freq, Then Lower Pressure/Mid-freq | Lower Pressure/Mid-freq, Then Higher Pressure/Variable-freq
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Half patients randomly assigned to HFCWC therapy first with a higher-pressure/variable frequency protocol. This entailed performing a 30 minute session with pressure of 10 and 5 minutes each at frequencies of 8,9, and 10 Hz followed by pressure of 6 and 5 minutes each at frequencies of 18, 19, and 20 Hz. This group subsequently crossed-over to the lower-pressure/mid-frequency HFCWC protocol after a washout period of 2 days. This entailed performing a HFCWC session using a pressure of 5 and frequency of 12 Hz for the entire 30 minute session. The other half of subjects were randomly assigned to perform the lower-pressure/mid-frequency protocol first followed by the higher pressure/mixed-frequency after the 2 day washout period
  VEST Airway Clearance System, Model 205 : Subjects will perform pulmonary function tests prior to and following each airway clearance therapy. All sputum produced during, and for 15 minutes following airway clearance therapy will be collected. Subjects
Arm/Group | All Study Participants
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Sputum Wet and Dry Weight
Description: All sputum expectorated during all HFCWC sessions was collected in a pre-weighed specimen container and immediately sealed. Half the subjects used higher pressure/mixed frequency on day 1 followed by lower pressure/mid-frequency on day 4. Half the patients performed lower pressure/mid-frequency on day 1 followed by higher pressure/mixed frequency on day 4. All specimens were immediately centrifuged at 21,150 g for 15 min at 4°C, and the supernatant was completely removed to eliminate saliva. The sputum "wet weight" was calculated after re-weighing the container with the sputum pellet. The container was then left open in an oven with the temperature set at 65°C for a minimum of 3 days to allow for complete desiccation. The sputum "dry weight" was calculated after re-weighing the container.
Time Frame: Produced during each airway clearance therapy session on days 1 and 4
Population: In a previous study with similar design,21 the standard deviation for the difference in the mean sputum wet weight between treatment arms was 4.6 g. Assuming the same standard deviation for the current study, enrollment of 16 subjects provided an 80% chance of detecting a 3.5-g difference in the sputum wet weights at a significance level of .05.
Measure: Median (Full Range); unit: grams
Groups:
- Sputum Wet Weight Higher Pressure/Variable Frequency; Sputum Wet Weight Lower Pressure/Mid-frequency: All sputum expectorated during all HFCWC sessions was collected in a pre-weighed specimen container and immediately sealed. Half the subjects used higher pressure/mixed frequency on day 1 followed by lower pressure/mid-frequency on day 4. Half the patients performed lower pressure/mid-frequency on day 1 followed by higher pressure/mixed frequency on day 4. All specimens were immediately centrifuged at 21,150 g for 15 min at 4°C, and the supernatant was completely removed to eliminate saliva. The sputum "wet weight" was calculated after re-weighing the container with the sputum pellet.
- Sputum Dry Weight Higher Pressure/Variable Frequency; Sputum Dry Weight Lower Pressure/Mid-frequency: All sputum expectorated during all HFCWC sessions was collected in a pre-weighed specimen container and immediately sealed. Half the subjects used higher pressure/mixed frequency on day 1 followed by lower pressure/mid-frequency on day 4. Half the patients performed lower pressure/mid-frequency on day 1 followed by higher pressure/mixed frequency on day 4. All specimens were immediately centrifuged at 21,150 g for 15 min at 4°C, and the supernatant was completely removed to eliminate saliva. The container was then left open in an oven with the temperature set at 65°C for a minimum of 3 days to allow for complete desiccation. The sputum "dry weight" was calculated after re-weighing the container.
Arm/Group | Sputum Wet Weight Higher Pressure/Variable Frequency | Sputum Wet Weight Lower Pressure/Mid-frequency | Sputum Dry Weight Higher Pressure/Variable Frequency | Sputum Dry Weight Lower Pressure/Mid-frequency
Number analyzed (Participants) | 16 | 16 | 16 | 15
grams | 6.4 [0.49 to 22.0] | 4.8 [0.24 to 15.0] | 0.20 [.009 to 0.62] | 0.12 [.0001 to 1.0]
Statistical Analysis 1: Comparison: Sputum Wet Weight Higher Pressure/Variable Frequency vs Sputum Wet Weight Lower Pressure/Mid-frequency vs Sputum Dry Weight Higher Pressure/Variable Frequency vs Sputum Dry Weight Lower Pressure/Mid-frequency; Test type: Superiority or Other; p = .02, ANCOVA; Mean Difference (Final Values) = .23, Standard Deviation .23

2. Secondary Outcome: Pre vs. Post Therapy Spirometry
Description: Spirometry was performed prior to, and immediately following, all HCWC sessions on Day 1. Spirometry was performed immediately prior to, and immediately following, all HFCWC sessions on Day 4. Spirometry was performed according to American Thoracic Society/European Respiratory Society standards.
Time Frame: Prior to and following each airway clearance therapy session on days 1 and 4
Population: Power calculation not performed for secondary outcomes.
Measure: Mean (Standard Deviation); unit: ml
Groups:
- Change in FEV1 Pre vs Post Higher Pressure/Variable Frequency; Change in FEV1 Pre vs Post Lower Pressure/Mid-frequency; Change in FVC Pre vs Post Higher Pressure/Variable Frequency; Change in FVC Pre vs Post Lower Pressure/Mid-frequency: Spirometry was performed prior to, and immediately following, all HCWC sessions on Day 1. Spirometry was performed immediately prior to, and immediately following, all HFCWC sessions on Day 4. Spirometry was performed according to American Thoracic Society/European Respiratory Society standards.
Arm/Group | Change in FEV1 Pre vs Post Higher Pressure/Variable Frequency | Change in FEV1 Pre vs Post Lower Pressure/Mid-frequency | Change in FVC Pre vs Post Higher Pressure/Variable Frequency | Change in FVC Pre vs Post Lower Pressure/Mid-frequency
Number analyzed (Participants) | 16 | 16 | 16 | 16
ml | 70 (90) | 90 (120) | 80 (160) | 80 (230)

3. Secondary Outcome: Rheology and in Vitro Cough Transportability of Sputum Produced Immediately Following Airway Clearance Therapy Session
Description: Sputum was collected during the 15 minutes immediately following HFCWC sessions on day 1 and day 4. Half the subjects performed higher-pressure/mixed frequency HFCWC on Day 1 followed by lower pressure/mid-frequency HFCWC on Day 4. The other half of subjects performed lower pressure/mid-frequency on Day 1 followed by higer pressure/mixed-frequency on Day 4. Samples were studied with a rheometer (AR1000, TA Instruments, New Castle, Delaware) to assess the dynamic frequency range of stress-strain of a 20 microliter sputum sample over driving frequencies of 1-100 rad/s. Shear storage modulus (G') and shear loss modulus (G") were determined from these curves after nondestructive creep transformation. G' (or dynamic elasticity) measures stored energy and is a property of ideal solids. G" is directly proportional to viscosity (viscosity x frequency) and is a property of ideal liquids.
Time Frame: Sputum produced during the 15 minutes immediately following airway clearance therapy sessions on day 1 and day 4
Population: power calculation not performed for secondary outcomes
Measure: Median (Full Range); unit: dynes/cm^2
Groups:
- G' Storage Modulus at 1 Rad/Sec Higher Pressure/Variable Freq; G' Storage Modulus at 1 Rad/Sec Lower Pressure/Mid-frequency; G' Storage Modulus 100 Rad/Sec Higher Pressure/Variable Freq; G' Storage Modulus 100 Rad/Sec Lower Pressure/Mid-frequency; G" Loss Modulus 1 Rad/Sec Higher Pressure/Variable Frequency; G" Loss Modulus 1 Rad/Sec Lower Pressure/Mid-frequency; G" Loss Modulus 100 Rad/Sec Higher Pressure/Variable Frequency; G" Loss Modulus 100 Rad/Sec Lower Pressure/Mid-frequency: Sputum was collected during the 15 minutes immediately following HFCWC sessions on day 1 and day 4. Half the subjects performed higher-pressure/mixed frequency HFCWC on Day 1 followed by lower pressure/mid-frequency HFCWC on Day 4. The other half of subjects performed lower pressure/mid-frequency on Day 1 followed by higer pressure/mixed-frequency on Day 4. Samples were studied with a rheometer (AR1000, TA Instruments, New Castle, Delaware) to assess the dynamic frequency range of stress-strain of a 20 microliter sputum sample over driving frequencies of 1-100 rad/s. Shear storage modulus (G') and shear loss modulus (G") were determined from these curves after nondestructive creep transformation. G' (or dynamic elasticity) measures stored energy and is a property of ideal solids. G" is directly proportional to viscosity (viscosity x frequency) and is a property of ideal liquids.
Arm/Group | G' Storage Modulus at 1 Rad/Sec Higher Pressure/Variable Freq | G' Storage Modulus at 1 Rad/Sec Lower Pressure/Mid-frequency | G' Storage Modulus 100 Rad/Sec Higher Pressure/Variable Freq | G' Storage Modulus 100 Rad/Sec Lower Pressure/Mid-frequency | G" Loss Modulus 1 Rad/Sec Higher Pressure/Variable Frequency | G" Loss Modulus 1 Rad/Sec Lower Pressure/Mid-frequency | G" Loss Modulus 100 Rad/Sec Higher Pressure/Variable Frequency | G" Loss Modulus 100 Rad/Sec Lower Pressure/Mid-frequency
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
dynes/cm^2 | 4.43 [0 to 162] | 4.61 [0 to 119] | 107.3 [11.2 to 1,352] | 130.7 [34 to 24,850] | 10.7 [0.4 to 205] | 7.4 [0.93 to 144] | 1,224 [383 to 11,270] | 862 [0 to 7,603]

4. Secondary Outcome: Patients' Perceived Comfort Using the Different Settings for the Vest Device
Description: Following each HFCWC session on day 1 and day 4, subjects completed a questionnaire that rated the comfort and efficacy of each HFCWC session using a 5-point scale. The questionnaire was entitled "Post-Therapy Questionnaire". Scale range for comfort ranged from 1 (very uncomfortable) to 3 (neutral) to 5 (very comfortable). Scale range for how "effective" the HFCWC session was ranged from 1 (minimally effective) to 3 (neutral) to 5 (very effective).
Time Frame: Immediately following each airway clearance therapy on day 1 and day 4
Population: power calculation not performed for secondary outcomes
Measure: Median (Full Range); unit: units on a scale
Groups:
- Perceived Comfort Higher Pressure/Variable Frequency; Perceived Comfort Lower Pressure/Mid-frequency: Following each HFCWC session on day 1 and day 4, subjects completed a questionnaire that rated the comfort of each HFCWC session using a 5-point scale. The questionnaire was entitled "Post-Therapy Questionnaire". Scale range for comfort ranged from 1 (very uncomfortable) to 3 (neutral) to 5 (very comfortable).
- Perceived Effectiveness Higher Pressure/Variable Frequency; Perceived Effectiveness Lower Pressure/Mid-frequency: Following each HFCWC session on day 1 and day 4, subjects completed a questionnaire that rated the comfort and efficacy of each HFCWC session using a 5-point scale. The questionnaire was entitled "Post-Therapy Questionnaire". Scale range for how "effective" the HFCWC session was ranged from 1 (minimally effective) to 3 (neutral) to 5 (very effective).
Arm/Group | Perceived Comfort Higher Pressure/Variable Frequency | Perceived Comfort Lower Pressure/Mid-frequency | Perceived Effectiveness Higher Pressure/Variable Frequency | Perceived Effectiveness Lower Pressure/Mid-frequency
Number analyzed (Participants) | 16 | 16 | 16 | 12
units on a scale | 4.5 [1 to 5] | 5 [1 to 5] | 4 [3 to 5] | 4 [3 to 5]

ADVERSE EVENTS:
Arm/Group | Lower Pressure/Mid-frequency | Higher Pressure/Variable Frequency
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

LIMITATIONS AND CAVEATS:
1. Sputum weights varied more than anticipated and the study was underpowered to detect differences in the primary outcomes.
2. Study not generalizable to patients that do not produce sputum or have an FEV1 < 40% predicted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No